CLINICAL TRIAL: NCT06877364
Title: Multicenter Phase I and II Clinical Study on Safety, Tolerability and Efficacy of GcMAF in Patients With Chronic Inflammatory Diseases
Brief Title: Safety, Tolerability and Efficacy of GcMAF in Patients With Chronic Inflammatory Diseases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW024
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Inflammation
Keywords: macrophages; inflamation regulation
MeSH Terms: conditions — Inflammation | interventions — vitamin D-binding protein-macrophage activating factor; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: GcMAF (Experimental): This arm includes patients receiving GcMAF at the recommended dose (determined in the open-label, dose-escalation Phase I portion of the study). GcMAF will be administered (e.g., subcutaneously) once or twice-weekly for approximately 12 - 16 weeks in the randomized Phase II portion. Efficacy will be measured using validated clinical scales (e.g., DAS28 for rheumatoid arthritis) and laboratory markers (CRP, ESR, etc.). Safety and tolerability will be monitored throughout the treatment period and in a follow-up phase (4 - 8 weeks).
  Interventions: Biological: GcMAF
- Placebo Comparator: Saline Injection (Placebo Comparator): This arm includes patients receiving a placebo injection (e.g., saline) under the same schedule (once or twice-weekly for 12-16 weeks) in the randomized Phase II portion of the study. Participants and investigators will be blinded to the treatment assignment. Clinical outcomes and safety profiles will be compared with those of the GcMAF arm to evaluate efficacy and confirm the overall safety of GcMAF.
  Interventions: Other: Placebo Injection (Saline)

INTERVENTIONS:
Biological: GcMAF — GcMAF is an immunomodulatory protein derived from vitamin D-binding protein via enzymatic deglycosylation. In this study, GcMAF will be administered (e.g., subcutaneously) once or twice-weekly for 12-16 weeks, followed by a 4-8-week observation period. The primary objectives include assessing clinical efficacy in chronic inflammatory conditions and confirming safety. GcMAF activates macrophages and dendritic cells, modulates M1/M2 profiles, and may reduce inflammatory markers such as CRP and ESR.
  Arms: Experimental: GcMAF
Other: Placebo Injection (Saline) — Participants in the placebo arm will receive a visually matching injection of normal saline (placebo) on the same schedule as the GcMAF arm (e.g., once or twice-weekly for 12-16 weeks). This allows for double-blind comparison of safety and efficacy endpoints. The placebo is designed to be identical in appearance and administration route to maintain blinding for investigators and participants.
  Arms: Placebo Comparator: Saline Injection

SUMMARY:
This study, titled "A Multicenter Phase I/II Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of GcMAF in Patients With Chronic Inflammatory Diseases" will investigate Gc Macrophage Activating Factor, a protein derived by enzymatic deglycosylation of vitamin D-binding protein. GcMAF activates macrophages and dendritic cells, modulates M1/M2 profiles, and shows anti-inflammatory effects. Phase I (open-label, dose-escalation) will assess safety, tolerability, and determine a Recommended Dose (RD). Phase II (randomized, double-blind, placebo-controlled) will evaluate efficacy and further confirm safety in a larger patient population with conditions such as moderate rheumatoid arthritis or chronic cystitis, refractory to standard therapies.

DETAILED DESCRIPTION:
This trial is designed to evaluate GcMAF, an immunomodulatory protein generated from vitamin D-binding protein (DBP) via specific enzymatic deglycosylation, in adults (≥18 years) with a confirmed chronic inflammatory disease (e.g., moderate rheumatoid arthritis, chronic cystitis) who have experienced inadequate response or intolerance to standard anti-inflammatory treatments (NSAIDs, corticosteroids, etc.). GcMAF's primary mechanism of action involves activating macrophages and dendritic cells, regulating cytokine production, and potentially offering anti-inflammatory as well as antitumor benefits, as indicated in preclinical studies on animal models with conditions such as adjuvant arthritis and hemorrhagic cystitis.

The study will be conducted in two phases. Phase I is an open-label, dose-escalation investigation comprising 3-4 cohorts receiving increasing doses of GcMAF (administered subcutaneously or intramuscularly). The primary objectives for Phase I are to determine the safety profile, tolerability, and maximum tolerated dose (MTD) or Recommended Dose (RD). This will involve continuous safety monitoring, assessment of adverse events (AEs) using CTCAE criteria, and evaluation of lab parameters (hematology, biochemistry, inflammatory markers). Secondary endpoints in Phase I include preliminary efficacy measures (changes in CRP, ESR, cytokines, and disease-activity scores) and (Cmax, Tmax, AUC, T½), along with possible measurement of antibodies to GcMAF.

Upon establishing the RD in Phase I, Phase II will be a randomized, double-blind, placebo-controlled trial enrolling approximately 60-120 patients. They will be allocated (1:1 or 1:1:1 if multiple GcMAF doses are tested) to receive either GcMAF (RD) or placebo for 12-16 weeks, followed by a 4-8-week observation period. The key inclusion criteria stipulate adult patients with documented chronic inflammatory disease and the ability to adhere to the protocol. Exclusion criteria include pregnancy or lactation, severe systemic illnesses (e.g., liver/kidney failure), active serious infections (HIV, TB, or active hepatitis B/C), recent participation in other experimental studies (<3 months), and hypersensitivity to protein products.

Phase II primary endpoints focus on clinical efficacy, measured by validated scores (e.g., DAS28 for rheumatoid arthritis, symptom indices for cystitis) and the proportion of patients achieving clinically significant improvement (e.g., DAS28 improvement ≥1.2 points). Secondary endpoints include ongoing safety assessments, laboratory markers of inflammation (CRP, ESR, cytokine profile), pharmacodynamic data (such as M1/M2 macrophage ratio), and patient-reported outcomes (e.g., SF-36, HAQ-DI). Statistical analyses will include descriptive methods in Phase I for safety and tolerability, and for Phase II comparative tests (t-test, ANOVA, or nonparametric equivalents) for continuous data and chi-square or Fisher's exact test for categorical response rates. Ultimately this trial seeks to confirm whether GcMAF offers a clinically meaningful reduction of inflammatory disease activity while maintaining an acceptable safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria
* Age ≥ 18 years, informed consent.
* Confirmed diagnosis of a chronic inflammatory disease (e.g., moderate rheumatoid arthritis or chronic cystitis, or another validated nosology) according to recognized criteria.
* Insufficient effect or intolerance of standard anti-inflammatory therapy (NSAIDs, GCS, etc.).
* Ability to comply with the study protocol.

Exclusion Criteria:

* Pregnancy, lactation (lack of safety data in this group).
* Severe systemic diseases (liver/renal failure, severe cardiovascular diseases, uncontrolled arterial hypertension).
* Active serious infections (HIV, tuberculosis, hepatitis B/C in the active phase).
* Previous participation in other experimental studies < 3 months ago.
* Severe allergy to protein components of the drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (Safety Assessment) | 4 weeks
  This outcome measures the incidence, severity, and type of treatment-emergent adverse events (AEs) associated with GcMAF administration, including any serious adverse events (SAEs). Adverse events will be graded using the Common Terminology Criteria for Adverse Events (CTCAE v5.0), which rates severity from Grade 1 (mild) to Grade 5 (death related to AE). A higher count of severe events indicates a worse safety profile.
Change in DAS28 Score | 16 Week
  The Disease Activity Score 28 (DAS28) is used to evaluate rheumatoid arthritis disease activity, though it can be adapted for other chronic inflammatory conditions as applicable. DAS28 ranges from 0.0 to 9.4, where higher scores indicate greater disease activity. A decrease in DAS28 score from baseline represents clinical improvement. For example, a DAS28 score under 2.6 is considered remission, while above 5.1 indicates high disease activity.

SECONDARY OUTCOMES:
Change in Serum C-Reactive Protein (CRP) | 16 weeks
  CRP is a laboratory measure of inflammation, reported in mg/L. Higher CRP values generally indicate more inflammation. This outcome will compare CRP levels at baseline versus the end of the active treatment period to assess the anti-inflammatory effect of GcMAF. A lower CRP at follow-up suggests improvement.
Change in Erythrocyte Sedimentation Rate (ESR) | 16 weeks
  ESR (mm/hr) is another indicator of systemic inflammation; higher values typically reflect more active inflammation. This outcome measure tracks the difference in ESR from baseline to post-treatment, allowing comparison between the GcMAF arm and placebo. A decrease in ESR indicates improvement.
Change in SF-36 Quality of Life Score | 16 weeks
  The 36-Item Short Form Survey (SF-36) measures overall health status across multiple domains (physical functioning, pain, vitality, mental health, etc.). Each domain is scored from 0 to 100, with higher scores indicating better health-related quality of life. The total SF-36 score is often reported as two main components (Physical and Mental), each ranging from 0 (worst) to 100 (best). An increase in SF-36 scores indicates an improvement in quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Center For New Medical Technologies, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No